CLINICAL TRIAL: NCT01645423
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-way Crossover Oral BE Study of Atorvastatin Ca 80 mg Tablets of Dr. Reddy's and Lipitor 80 mg Tablets of Pfizer in Healthy Adult, Human Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Atorvastatin Calcium Tablets, 80 mg of Dr. Reddy's Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 09-VIN-105
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Bioequivalence; Atorvastatin calcium; crossover
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin Calcium Tablets, 80 mg (Experimental): Atorvastatin Calcium Tablets, 80 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Atorvastatin Calcium Tablets, 80 mg
- Lipitor 80 mg Tablets (Active Comparator): Lipitor 80 mg Tablets of Pfizer Ireland Pharmaceuticals
  Interventions: Drug: Atorvastatin Calcium Tablets, 80 mg

INTERVENTIONS:
Drug: Atorvastatin Calcium Tablets, 80 mg — Atorvastatin Calcium Tablets, 80 of Dr. Reddy's Laboratories Limited
  Other Names: Lipitor 80 mg Tablets

SUMMARY:
The purpose of this study is to compare and evaluate the single-dose oral bioavailability and to monitor the safety of subjects.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two-way crossover oral bioequivalence' study of Atorvastatin Calcium 80 mg Tablets of Dr. Reddy's and Lipitor 80 mg Tablets of Pfizer Ireland Pharmaceuticals in healthy adult, human subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 45 years (both inclusive).
2. Subjects' weight within normal range according to normal values for Body Mass Index (1 8.5 to 24.9 kg/m2) with minimum of 50 kg weight.
3. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations (Annexure IIIa) within the clinically acceptable reference range (Annexure IIIb).
4. Subjects having normal 12-lead electrocardiogram (ECG).
5. Subjects having normal chest X-Ray (P/A view) whose X-Ray was taken not more than 6 months prior to the dosing of Period 0 1.
6. Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
7. Subjects having negative alcohol breath test.
8. Subjects willing to adhere to the protocol requirements and to provide written informed consent.

Exclusion Criteria:

Subjects will be excluded from the study, if they meet any of the following criteria:

1. Hypersensitivity to Atorvastatin or related class of drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
3. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 1 month of the study starting.
4. History or presence of significant alcoholism or drug abuse in the past one year.
5. History or presence of significant smoking (more than 10 cigarettes or beedi's/day).
6. History or presence of asthma, urticaria or other significant allergic reactions.
7. History or presence of significant gastric andlor duodenal ulceration.
8. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
9. History or presence of cancer.
10. Difficulty with donating blood.
11. Difficulty in swallowing solids like tablets or capsules.
12. Use of any prescribed or OTC medication during last two weeks prior to dosing in period 0 1.
13. Major illness during 3 months before screening.
14. Participation in a drug research study within past 3 months.
15. Donation of blood in the past 3 months before screening.
16. Consumption of grapefruit juice, xanthine-containing products, tobacco containing products or alcohol for within 48 hours prior to dosing.
17. Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
18. History or presence of significant easy bruising or bleeding.
19. History or presence of significant recent trauma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | Pre-dose at 0.00 hour and post-dose at 0.25, 0.50, 0.75, 1.00, 1.25, 1.50 1.75, 2.00, 2.25,2.50, 2.75, 3.00, 3.33, 3.67,4.00,4.50, 5.00,6.00, 8.00, 10.00, 12.00, 16.00,24.00, 36.00, 48.00 and 72.00 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dharmesh Domadia, MD, Principal Investigator — Veeda Clinical Research Pvt. Ltd.,
Locations (1):
- Veeda Clinical Research Pvt. Ltd.,, Ahmedabad, Gujarat, India